CLINICAL TRIAL: NCT04913987
Title: PPK: A Functional and Clinical Comparison of a Partial and Total Knee Replacement
Brief Title: Persona Partial Knee Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ortho 18-03
Record Dates: First submitted 2019-07-17; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Total knee arthroplasty; Partial knee arthroplasty; Unicondylar knee arthroplasty; Randomised controlled trial; Functional biomechanical assessment; Movement analysis; Gait analysis

STUDY DESIGN:
Intervention Model Description: Consecutive patients placed in to one of two groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total knee (Experimental): Standard care
  Interventions: Device: Stryker Triathlon total knee replacement
- Partial knee (Experimental): Intervention using relatively new partial knee.
  Interventions: Device: Zimmer Biomet Persona Partial Knee unicondylar knee replacement

INTERVENTIONS:
Device: Stryker Triathlon total knee replacement — Knee arthroplasty using a standard care total knee.
  Arms: Total knee
Device: Zimmer Biomet Persona Partial Knee unicondylar knee replacement — Knee arthroplasty using the Zimmer Biomet Persona Partial Knee (PPK).
  Other Names: Zimmer Biomet Persona Partial Knee (PPK)
  Arms: Partial knee

SUMMARY:
This study will compare functional and clinical outcomes of partial knee joint replacement using the Persona Partial Knee (PPK) and a standard care total knee replacement. Reported benefits of unicompartmental knee arthroplasty (UKA) compared to total knee arthroplasty (TKA) are less invasive surgery, less post-operative pain, quicker recovery, shorter inpatient stay, preservation of the anterior cruciate ligament (ACL), better knee function and lower risk of complications. Also, the PPK more closely matches the anatomy of knee and has more sizing options. These aim to allow the surgeon to reconstruct the knee to better match the native knee and achieve natural function.

Little data exists which investigates biomechanical function of patients after UKA or comparisons between UKA and TKA and none investigating the PPK. Available data focuses on level walking which is not particularly challenging for these patients and is unlikely to highlight biomechanical differences between UKA and TKA. The investigators will investigate biomechanical differences between UKA and TKA during more challenging activities. These will mirror activities of everyday life: sitting into/rising from a chair, stepping, walking on a slope.

The investigators will investigate level walking as all studies of this nature report these data. Unlike TKA, UKA retains the ACL. The soft tissues of the knee play a role in balance control and the investigators will assess this with single leg balancing. Biomechanical differences will be assessed using 3D motion analysis before and after surgery (6 and 12 months). Comparisons will be made within and between groups and between the patient groups and existing healthy data. Radiographic and patient reported outcomes (satisfaction, pain and functional abilities) will be investigated.

Fifty patients will be recruited and randomised to undergo TKA or UKA. Only patients who are suitable for UKA will be recruited. Data for 25 healthy, matched controls from the investigator's existing healthy control database will be extracted.

DETAILED DESCRIPTION:
All patients identified as possible participants for the study will be given a "consent to be approached for research" form on arrival at the clinic by the unit co-ordinator. On this, patients can indicate their willingness or otherwise to have the study explained to them. The completed form will be given to their consultant prior to their appointment. Patients who have indicated willingness, and who are deemed suitable for the study following the consultation, will have the study introduced to them by their consultant, who will then ask a member of the research team to fully explain the study. These patients will be given a copy of the Participant Information Sheet (PIS) to take away.

At a later date (at least a day after receiving the PIS), these patients will be contacted by telephone to ask for verbal consent. Patients will also have the opportunity to ask questions about the study. Verbal consent will not be binding, but is necessary to give the research team time to arrange pre-operative study interventions. Written consent will be taken when the patient arrives for the pre-operative biomechanical testing session, once the researcher is happy that the patient is fully informed. Consent will be sought by the principal investigator or one of his delegates.

Standard care for knee arthroplasty patients at the GJNH has them completing the Oxford Knee Score (OKS) and the EQ-5D pre-operatively and at six weeks post-operatively. In addition, satisfaction is measured on a five point Likert scale six weeks post-operatively. Study participants will also be asked to complete these three measures at six and 12 months post-operatively. Two additional questionnaires will be used in the study. The UCLA Activity Score will be used pre-operatively and at six weeks, six months and 12 months post-operatively. The Forgotten Joint Score (FJS) will be used at the three post-operative time points (six week, six months and 12 months).

At 12 months post-operatively, study participants will have two radiographs taken (short AP and lateral views) which are additional to the standard care radiography protocol. The six and 12 month post-operative visits are additional to standard care and, as such, participants will be offered the reimbursement of reasonable travelling costs. Biomechanical assessment using clinical movement analysis (CMA) in the movement analysis laboratory (MAL) at the GJNH will be carried out on three occasions (pre-operatively and at six and 12 months post-operatively). The MAL is a purpose built facility with restricted access for privacy. Changing facilities are provided within the laboratory for participants to change from their outdoor clothes into a T-shirt and shorts for the testing. They will also be asked to perform the testing barefoot. At this point a health care support worker will apply a bandage to the operated knee covering the wound to maintain the blinding of the person collecting the biomechanical data. During these assessments, participants will have a number of small reflective markers attached to their body using toupé tape. The movements of these markers will be tracked by a number of infrared cameras connected to a computer. The data collected in this manner can generate dynamic angles of the joints during the study tasks. In addition, force plates embedded in the floor will measure forces generated during the study tasks which can be converted to forces at each of the joints. During the assessment, participants will be asked to perform a number of activities of daily living; level walking, incline and decline walking, stand-to-sit-to-stand, step ascent and descent and single leg balance. Participants will be asked to perform each task a minimum of three times to ensure that three representative samples of each task are obtained; except for the single leg balance, which will be performed once for each limb. Pre-operative testing will determine baseline function while post-operative assessment will highlight any changes in function.

Following recruitment, participants will be randomised to receive the PPK unicondylar knee implant or the total kneeimplant routinely used in the GJNH. Surgery will be performed as per the surgeons' standard practice using the implant the participant was randomised to receive. After their 12 months follow-up, the participants' involvement in the study will be over.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for medial unicompartmental knee arthroplasty
* Aged between 18 and 75 years inclusive
* Taller than 1.5m in height (the 10th percentile for the population)
* Functionally intact anterior cruciate ligament
* Able to give informed consent
* Able to return to GJNH for follow-up
* BMI under 40

Exclusion Criteria:

* Inflammatory joint disease e.g. rheumatoid arthritis
* Previous hip procedure in the previous twelve months
* Previous knee surgery other than arthroscopy and medial menisectomy
* Previous ankle surgery
* Symptomatic foot, hip or spinal pathology
* Any medical condition limiting normal ambulation e.g. stroke, Charcot-Marie-Tooth disease, severe lymphedema, advanced cardiac disease
* Unable to read and understand English and follow verbal and visual instructions unless they can bring a relative or friend to all study assessments to act as a translator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Knee flexion | 12 months post-operatively
  Maximum knee flexion in degrees during step descent measured using movement analysis

SECONDARY OUTCOMES:
Radiographic assessment of component/bone interface stability | 12 months post-operatively
  Component position, orientation and signs of loosening using a modified Knee Society Radiographic Assessment Tool (No score produced)
Survivorship | 12 months
  Number of implants in situ
Patient satisfaction: 5 point Likert scale | 12 months post-operatively
  Patient satisfaction on a 5 point Likert scale ( Very satisfied, Satisfied, Unsure, Dissatisfied, Very dissatisfied)

OTHER OUTCOMES:
Patient reported outcome (Oxford Knee Score) | 12 months post-operatively
  Patient pain and function measured using the Oxford Knee Score questionnaire (12 to 60, best to worst outcome)
Patient reported outcome (EuroQual 5D-5L questionnaire) | 12 months post-operatively
  Change in overall health compared to pre-operatively (Positive change is an improvement. Reported as a weighted index score where max is 1 and min is based on national data)
Patient reported outcome (Forgotten Joint Score) | 12 months post-operatively
  Patient awareness of their replacement knee using the Forgotten Joint Score (0-100, poor to good outcome)
Patient reported outcome (University of California Los Angelees Activity Score) | 12 months post-operatively
  Patient activity level measured using the UCLA Activity Score (10 item activity grade from worst to best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Nichoas Ohlyl, FRCS Ed, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sculco TP. Orthopaedic crossfire--can we justify unicondylar arthroplasty as a temporizing procedure? in opposition. J Arthroplasty. 2002 Jun;17(4 Suppl 1):56-8. doi: 10.1054/arth.2002.32687. PMID 12068406
- [Background] Deshmukh RV, Scott RD. Unicompartmental knee arthroplasty: long-term results. Clin Orthop Relat Res. 2001 Nov;(392):272-8. PMID 11716395
- [Background] Alnachoukati OK, Barrington JW, Berend KR, Kolczun MC, Emerson RH, Lombardi AV Jr, Mauerhan DR. Eight Hundred Twenty-Five Medial Mobile-Bearing Unicompartmental Knee Arthroplasties: The First 10-Year US Multi-Center Survival Analysis. J Arthroplasty. 2018 Mar;33(3):677-683. doi: 10.1016/j.arth.2017.10.015. Epub 2017 Oct 16. PMID 29113757
- [Background] Forster-Horvath C, Artz N, Hassaballa MA, Robinson JR, Porteous AJ, Murray JR, Newman JH. Survivorship and clinical outcome of the minimally invasive Uniglide medial fixed bearing, all-polyethylene tibia, unicompartmental knee arthroplasty at a mean follow-up of 7.3years. Knee. 2016 Dec;23(6):981-986. doi: 10.1016/j.knee.2016.07.003. Epub 2016 Aug 6. PMID 27506988
- [Background] Braito M, Giesinger JM, Fischler S, Koller A, Niederseer D, Liebensteiner MC. Knee Extensor Strength and Gait Characteristics After Minimally Invasive Unicondylar Knee Arthroplasty vs Minimally Invasive Total Knee Arthroplasty: A Nonrandomized Controlled Trial. J Arthroplasty. 2016 Aug;31(8):1711-6. doi: 10.1016/j.arth.2016.01.045. Epub 2016 Feb 10. PMID 26979765
- [Background] Liddle AD, Judge A, Pandit H, Murray DW. Adverse outcomes after total and unicompartmental knee replacement in 101,330 matched patients: a study of data from the National Joint Registry for England and Wales. Lancet. 2014 Oct 18;384(9952):1437-45. doi: 10.1016/S0140-6736(14)60419-0. PMID 25012116
- [Background] Svard UC, Price AJ. Oxford medial unicompartmental knee arthroplasty. A survival analysis of an independent series. J Bone Joint Surg Br. 2001 Mar;83(2):191-4. doi: 10.1302/0301-620x.83b2.10966. PMID 11284563
- [Background] Goodfellow J, O'Connor J. The anterior cruciate ligament in knee arthroplasty. A risk-factor with unconstrained meniscal prostheses. Clin Orthop Relat Res. 1992 Mar;(276):245-52. PMID 1537161
- [Background] Deschamps G, Lapeyre B. [Rupture of the anterior cruciate ligament: a frequently unrecognized cause of failure of unicompartmental knee prostheses. Apropos of a series of 79 Lotus prostheses with a follow-up of more than 5 years]. Rev Chir Orthop Reparatrice Appar Mot. 1987;73(7):544-51. French. PMID 3438510
- [Background] Banks SA, Fregly BJ, Boniforti F, Reinschmidt C, Romagnoli S. Comparing in vivo kinematics of unicondylar and bi-unicondylar knee replacements. Knee Surg Sports Traumatol Arthrosc. 2005 Oct;13(7):551-6. doi: 10.1007/s00167-004-0565-x. Epub 2005 Jan 20. PMID 15660274
- [Background] Andriacchi TP, Galante JO, Fermier RW. The influence of total knee-replacement design on walking and stair-climbing. J Bone Joint Surg Am. 1982 Dec;64(9):1328-35. No abstract available. PMID 7142241
- [Background] Komnik I, Peters M, Funken J, David S, Weiss S, Potthast W. Non-Sagittal Knee Joint Kinematics and Kinetics during Gait on Level and Sloped Grounds with Unicompartmental and Total Knee Arthroplasty Patients. PLoS One. 2016 Dec 21;11(12):e0168566. doi: 10.1371/journal.pone.0168566. eCollection 2016. PMID 28002437
- [Background] Komnik I, Weiss S, Fantini Pagani CH, Potthast W. Motion analysis of patients after knee arthroplasty during activities of daily living--a systematic review. Gait Posture. 2015 Feb;41(2):370-7. doi: 10.1016/j.gaitpost.2015.01.019. Epub 2015 Jan 28. PMID 25680471
- [Background] Jones GG, Kotti M, Wiik AV, Collins R, Brevadt MJ, Strachan RK, Cobb JP. Gait comparison of unicompartmental and total knee arthroplasties with healthy controls. Bone Joint J. 2016 Oct;98-B(10 Supple B):16-21. doi: 10.1302/0301-620X.98B10.BJJ.2016.0473.R1. PMID 27694511
- [Background] Wiik AV, Aqil A, Tankard S, Amis AA, Cobb JP. Downhill walking gait pattern discriminates between types of knee arthroplasty: improved physiological knee functionality in UKA versus TKA. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1748-55. doi: 10.1007/s00167-014-3240-x. Epub 2014 Aug 27. PMID 25160471
- [Background] Fu YC, Simpson KJ, Brown C, Kinsey TL, Mahoney OM. Knee moments after unicompartmental knee arthroplasty during stair ascent. Clin Orthop Relat Res. 2014 Jan;472(1):78-85. doi: 10.1007/s11999-013-3128-y. PMID 23836240
- [Background] Shankar S, Tetreault MW, Jegier BJ, Andersson GB, Della Valle CJ. A cost comparison of unicompartmental and total knee arthroplasty. Knee. 2016 Dec;23(6):1016-1019. doi: 10.1016/j.knee.2015.11.012. Epub 2016 Oct 31. PMID 27810433
- [Background] Willis-Owen CA, Brust K, Alsop H, Miraldo M, Cobb JP. Unicondylar knee arthroplasty in the UK National Health Service: an analysis of candidacy, outcome and cost efficacy. Knee. 2009 Dec;16(6):473-8. doi: 10.1016/j.knee.2009.04.006. Epub 2009 May 22. PMID 19464898
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Fenner VU, Behrend H, Kuster MS. Joint Mechanics After Total Knee Arthroplasty While Descending Stairs. J Arthroplasty. 2017 Feb;32(2):575-580. doi: 10.1016/j.arth.2016.07.035. Epub 2016 Aug 13. PMID 27642045